CLINICAL TRIAL: NCT05811312
Title: Brain Connectivity Changes With Spinal Cord Stimulation Treatment of Chronic Pain: A Resting State NIRS/EEG Study
Brief Title: Brain Connectivity Changes With Spinal Cord Stimulation and Treatment of Chronic Pain: A Resting State NIRS/EEG Study
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F4389-P
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain
Keywords: chronic pain; neuropathic pain; spinal cord stimulation; fNIRS; electroencephalography
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — fNIRS/EEG, Numeric pain rating scale, EQ-5D-5L, Patients Global Impression of Change, PROMIS-29 Profile v2.1, PainDetect and Actigraphy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1-individuals who are naïve to SCS: Individuals with chronic neuropathic pain who are naïve to SCS and were selected for SCS trial period as part of their clinical care will participate in two study visits: before the beginning of the SCS trial and the end of the trial period. Data collection will be consistent across all data collection timepoints (T1 - T3) and include rs-fNIRS/EEG and clinical pain measures.
- Cohort 2-individuals with effective implanted SCS 6 months: Cohort 2: Participants with effective implanted SCS 6 months will participate in three study visits conducted 24-48 hours apart. Data will be collected during SCS use and following an SCS washout period. Data collection will be consistent across all data collection timepoints(T1-T4) and include rs-fNIRS/EEG and clinical pain measures. Both cohorts will receive paresthesia based SCS.

SUMMARY:
This study aims to assess how use of spinal cord stimulation for the treatment of chronic pain impacts brain structure and function. The investigators will use a non-invasive neuroimaging technique called resting state Near Infrared Spectroscopy and Electroencephalography (rs-fNIRS/EEG). The investigators will enroll Veterans who are currently receiving care at the Medical Center and who are either long term users of SCS for the treatment of their chronic pain or being evaluated for use of SCS to treat their pain.

DETAILED DESCRIPTION:
Chronic pain is a complex neurological disease that adversely impacts function and quality of life. Brain structure and function are altered when an individual is in the chronic pain state. Furthermore, chronic pain is associated with disruptions in functional brain connectivity. Spinal cord stimulation (SCS) is a clinically available non-pharmacological therapy that is used in the management of chronic pain. Although SCS is effective for many, there are individuals who do not benefit. Therefore, in order to better understand brain mechanisms that underlie SCS treatment of chronic pain and to develop brain biomarkers of SCS efficacy, the investigators propose to evaluate functional brain changes in response to SCS. Finding a brain signature of pain relief in response to SCS would improve understanding of how SCS alleviates chronic pain and may help to identify those most likely to respond. The main objective of this study is to assess changes in brain connectivity in response to SCS in individuals with chronic neuropathic pain. The investigators will study two cohorts: Cohort 1 - naïve to SCS patients who are undergoing SCS trial period; Cohort 1 - long-term SCS users ( 6 months post implantation). The investigators aim to identify neurophysiological brain signatures of pain relief in these two populations using resting state Near Infrared Spectroscopy and Electroencephalography (rs-fNIRS/EEG). Study Design: The investigators will enroll Veterans with refractory chronic neuropathic pain who are currently receiving clinical care within the medical center. Cohort 1: Individuals with chronic neuropathic pain who are naïve to SCS and were selected for SCS trial period as part of their clinical care will participate in two study visits: before the beginning of the SCS trial and the end of the trial period. Data collection will be consistent across all data collection timepoints (T1 - T3) and include rs-fNIRS/EEG and clinical pain measures. Cohort 2: Participants with effective implanted SCS 6 months will participate in three study visits conducted 24-48 hours apart. Data will be collected during SCS use and following an SCS washout period. Data collection will be consistent across all data collection timepoints(T1-T4) and include rs-fNIRS/EEG and clinical pain measures. Both cohorts will receive paresthesia based SCS. AIM 1 is to characterize neurophysiological (rs-fNIRS/EEG) brain signature of pain relief during the SCS trial period for patients with chronic neuropathic pain who are naïve to SCS. AIM 2 is to characterize neurophysiological (rs-fNIRS/EEG) brain signature of pain relief in patients with chronic neuropathic pain who have utilized SCS for 6 months. Outcome Measures to address both aims include rs-functional connectivity (rs-fNIRS/EEG); and a composite clinical pain assessment that will include Numeric Pain Rating Scale (NPRS), Patient Reported Outcomes Measurement Information System-29 profile v2.1(PROMIS-29); EQ-5D-5L; Patient Global Impression of Change (PGIC); painDetect; and activity monitoring. Significance: Studying changes in brain connectivity in response to SCS will provide insight into the treatment mechanism of SCS. Use of neuroimaging methods such as rs-fNIRS/EEG that can be easily applied in the clinical setting to further refine patient selection for SCS may improve outcome in SCS therapy. This grant will provide preliminary data for future studies aimed at developing biomarkers of pain-relief with SCS treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and a US veteran
* Diagnosis of chronic neuropathic pain.
* Current patient at Cleveland VA Medical Center receiving care via Pain Medicine Center.
* Current user of tonic parasthesia-based SCS (pain relief 50% according to NPRS) or undergoing trial SCS period as part of clinical care.
* Able to provide informed consent.
* Medically and psychologically stable.

Exclusion Criteria:

* Metal in the skull or deformity of the skull
* Pregnancy or pregnancy planning during the study period.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with chronic pain who are being treated as part of their clinical care with spinal cord stimulation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in resting state Functional Connectivity | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  resting state functional connectivity will be evaluated with fNIRS and EEG. We will model "response to SCS" with changes in resting state functional connectivity between five bilateral cortical regions. These regions are the medial prefrontal cortex (mPF), dorsolateral prefrontal cortex (DLPFC), primary motor cortex (M1), primary sensory cortex (S1), and posterior parietal cortex (PPC). Brain connectivity will be evaluated with fNIRS and EEG. Prefrontal medial cortex and posterior temporoparietal regions are good proxy measures of DMN activity using fNIRS.45-47 DMN nodes include additional deep brain structures18 but they are outside the field of view for most fNIRS instruments. We will evaluate S1 for its role in pain processing, M1 for its contribution to pain sensation via thalamic inhibition, and DLPFC for its known role in cognitive and affective pain processing.
Change in Numeric pain rating scale | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  NPRS measures pain intensity. Individuals select a number on a 0-10 scale that best describes the intensity of their current, best and worst pain levels; 0-10 scale, with 10 indicating maximum pain.

SECONDARY OUTCOMES:
Change in EQ-5D-5L | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  EQ-5D-5L is a 5-domain health-related quality of life measure; -0.59-1.00 scale, with 1=best health state.
Change in Patients Global Impression of Change (PGIC) | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  Patient's Global Impression of Change (PGIC) is a 7-point scale to assess patient perception of change in response to treatment. 1=no change, and 7=a great deal better.
Change in PROMIS-29 Profile v2.1 | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  PROMIS-29 Profile v2.1 is a questionnaire covering 7 domains including physical function, anxiety, depression, fatigue, sleep disturbance, participation in social roles/activities, and pain interference. Higher T-scores indicate more severity/worse health.
Change in PainDetect | Cohort 1: day 1 and between days 5-9; Cohort 2: day 1 and between days 3-6
  PainDetect is a self-report measure that was developed to assess neuropathic pain in adults with low back pain; 0-38 points, with higher score more indicative of neuropathic pain.
Change in Actigraphy | Cohort 1-between 5 and 9 days; Cohort 2-between 3-6 days.
  Activity monitoring using a wrist-worn device (Actigraphy) will be utilized to monitor real-life activity and sleep patterns; calculating % time active versus sedentary.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Pundik, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No